CLINICAL TRIAL: NCT00759902
Title: A Randomized Two-way Crossover, Single-Dose, Open-Label Study to Evaluate the Bioequivalence of a Test Formulation of KADIAN (2 x 10mg) Capsules Compared to a KADIAN 20 mg Capsule in Healthy Adult Subjects Under Fasted Conditions
Brief Title: Comparison of Two KADIAN 10 mg Capsules to a KADIAN 20 mg Capsule Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-073-SA
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2009-09-01 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: bioequivalence; 10 mg; KADIAN capsules; 20 mg; under fasted conditions
MeSH Terms: interventions — Morphine; Capsules

ARMS (2):
- 1 (Other): Treatment A (test product) followed by Treatment B (reference product)
  Interventions: Drug: morphine sulfate extended-release capsules; Drug: KADIAN (morphine sulfate extended-release) capsules
- 2 (Other): Treatment B (reference product) followed by Treatment A (test product)
  Interventions: Drug: morphine sulfate extended-release capsules; Drug: KADIAN (morphine sulfate extended-release) capsules

INTERVENTIONS:
Drug: morphine sulfate extended-release capsules — 2 x 10 mg, single-dose capsule
  Other Names: Treatment A; Test product
Drug: KADIAN (morphine sulfate extended-release) capsules — 1 x 20 mg, single-dose capsule
  Other Names: Treatment B; Reference product

SUMMARY:
The objective of this single-dose, open-label, randomized, two-treatment, two-period crossover study was to compare the relative bioavailability of a test formulation of KADIAN (2 x 10 mg) capsules manufactured by Alpharma Inc. to an equivalent oral dose of the commercially available reference product, KADIAN (1 x 20 mg)capsules manufactured by Alpharma Branded Products Inc. following an overnight fast of at least 10 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a male or non-pregnant, non-breast-feeding female.
* Subject must be between 18 and 55 years of age (inclusive).
* Subject's Body Mass Index (BMI) must be between 18 and 30 kg/m2 (inclusive), and subject must weigh a minimum of 50 kg (110 lbs).
* Female subjects - not surgically sterile or at least two years postmenopausal - must agree to utilize one of the following forms of contraception, if sexually active with a male partner, at least from screening through completion of the study. Approved forms of contraception are abstinence, hormonal (oral, implant, transdermal or injection) in use at least 3 consecutive months prior to first dose of study medication, double barrier (condom and diaphragm with spermicide), intra-uterine device (IUD), or vasectomized partner (6 months minimum since vasectomy).
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to completion of any study-specific procedures.
* Subject is willing and able to remain in the study unit for the entire duration of each confinement period and return to the study site for all outpatient visits.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic or psychiatric disease or any other condition which, in the opinion of the Investigator would jeopardize the safety of the subject or the validity of the study results.
* Has a clinically significant abnormal finding on the physical exam, medical history, ECG or clinical laboratory results at screening.
* History or presence of allergic or adverse response to the KADIAN or related drugs.
* Has been on a significantly abnormal diet during the four weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in another clinical trial within 30 days prior to first dose of study medication.
* Has used any over-the-counter (OTC) medication including nutritional supplements, within 7 days prior to the first dose of study medication.
* Has used any prescription medication, except hormonal contraceptive or hormonal replacement therapy, within 14 days prior to the first dose of study medication.
* Has been treated with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication.
* Has smoked or used tobacco products within 60 days prior to the first dose of study medication.
* Has a history of treatment for substance abuse (including alcohol) in the past 5 years.
* Is a female with a positive pregnancy test result.
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates).
* Has had a positive test for, or has been treated for Hepatitis B, Hepatitis C or HIV.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P. Doherty, DO, Principal Investigator — CEDRA Clinical Research, LLC
Locations (1):
- CEDRA Clinical Research, LLC, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1: Treatment A or B: Treatment A (test product) followed by Treatment B (reference product)
- Period 2: Treatment A or B: Treatment B (reference product) followed by Treatment A (test product)
Period: Overall Study
Arm/Group | Period 1: Treatment A or B | Period 2: Treatment A or B
Started | 18 | 18
Completed | 18 | 17
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1: Treatment A or B | Period 2: Treatment A or B | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.6 (9.6) | 31.7 (8.9) | 31.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Morphine Concentration
Time Frame: 0 (predose), and 2,4,6,6.5,7,7.5,8,8.5,9,9.5,10,12,18,24,30,36,48 hrs
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- KADIAN 10 mg Capsules: 2 x 10 mg KADIAN capsules
- KADIAN 20 mg Capsules: 1 x 20 mg KADIAN capsules
Arm/Group | KADIAN 10 mg Capsules | KADIAN 20 mg Capsules
Number analyzed (Participants) | 35 | 35
ng/mL | 5.23 (2.01) | 4.15 (1.35)
Statistical Analysis 1: Comparison: KADIAN 10 mg Capsules vs KADIAN 20 mg Capsules; Test type: Non-Inferiority or Equivalence — The 90% confidence intervals for the ratios (test/reference) of the least squares means of the non-transformed parameters Cmax, AUClast, AUCinf, Tmax, λz, and T1/2, were calculated; ANOVA; log-transformation; mean ratio = 123.0, 90% CI [112.9 to 134.1]

2. Secondary Outcome: Time of Maximum Plasma Morphine Concentration
Time Frame: 0 (predose), and 2,4,6,6.5,7,7.5,8,8.5,9,9.5,10,12,18,24,30,36,48 hrs
Measure: Median (Full Range); unit: hr
Arm/Group | KADIAN 10 mg Capsules | KADIAN 20 mg Capsules
Number analyzed (Participants) | 35 | 35
hr | 7.50 (2.15) [6.00 to 12.00] | 7.50 (3.82) [6.00 to 18.00]

3. Secondary Outcome: Area Under the Curve to the Last Measurable Time Point for Plasma Morphine
Time Frame: 0 (predose), and 2,4,6,6.5,7,7.5,8,8.5,9,9.5,10,12,18,24,30,36,48 hrs
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | KADIAN 10 mg Capsules | KADIAN 20 mg Capsules
Number analyzed (Participants) | 35 | 35
hr*ng/mL | 84.45 (22.29) | 82.94 (21.01)
Statistical Analysis 1: Comparison: KADIAN 10 mg Capsules vs KADIAN 20 mg Capsules; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; log-transformation; mean ratio = 101.7, 90% CI [98.5 to 104.9]

4. Secondary Outcome: Area Under the Curve to Infinity for Plasma Morphine
Time Frame: 0 (predose), and 2,4,6,6.5,7,7.5,8,8.5,9,9.5,10,12,18,24,30,36,48 hrs
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | KADIAN 10 mg Capsules | KADIAN 20 mg Capsules
Number analyzed (Participants) | 31 | 33
hr*ng/mL | 102.1 (31.63) | 100.0 (28.52)
Statistical Analysis 1: Comparison: KADIAN 10 mg Capsules vs KADIAN 20 mg Capsules; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; log-transformation; mean ratio = 102.9, 90% CI [99.3 to 106.5]

ADVERSE EVENTS:
Arm/Group | Arm 1: Treatment A Followed by Treatment B | Arm 2: Treatment B Followed by Treatment A
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 10 | 10
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Arm 1: Treatment A Followed by Treatment B | Arm 2: Treatment B Followed by Treatment A
Headache (Nervous system disorders) | 3/18 (3) | 6/18 (6)
Nausea (Gastrointestinal disorders) | 4/18 (4) | 3/18 (3)
Bowel (Gastrointestinal disorders) | 1/18 (1) | 1/18 (1)
Chest Pain (Cardiac disorders) | 1/18 (1) | 0/18 (0)
Constipation (Gastrointestinal disorders) | 2/18 (2) | 0/18 (0)
Flatulence (Gastrointestinal disorders) | 1/18 (1) | 0/18 (0)
Abdominal Pain (Gastrointestinal disorders) | 1/18 (1) | 2/18 (2)
Dizziness (Nervous system disorders) | 1/18 (1) | 1/18 (1)
Paraesthesia (Nervous system disorders) | 1/18 (1) | 0/18 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1/18 (1) | 0/18 (0)
Palpitations (Cardiac disorders) | 1/18 (1) | 0/18 (0)
Abnormal Dreams (Psychiatric disorders) | 0/18 (0) | 1/18 (2)
Skin Laceration (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/18 (1)
Vomiting (Gastrointestinal disorders) | 0/18 (0) | 1/18 (1)
Genital Herpes (Infections and infestations) | 0/18 (0) | 1/18 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0/18 (0) | 1/18 (1)
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/18 (1)
Hunger (General disorders) | 0/18 (0) | 1/18 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 0/18 (0) | 1/18 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No